CLINICAL TRIAL: NCT01922557
Title: The Association of Thoracic Fluid Content and Acute Lung Injury in Liver Transplantation
Brief Title: Thoracic Fluid Content and Acute Lung Injury
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201012081RC
Record Dates: First submitted 2013-07-11; First posted 2013-08-14 (Estimated); Last update posted 2013-08-14 (Estimated); Status verified 2013-08

CONDITIONS: Acute Lung Injury
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (1):
- NICOM
  Interventions: Device: NICOM

INTERVENTIONS:
Device: NICOM — NICOM monitoring thoracic fluid content at baseline(T1), anhepatic phase(T2), 30 mins after reperfusion(T3) and 2 hrs after reperfusion(T4).

SUMMARY:
To study the association of the thoracic fluid content and acute lung injury during liver transplantation.

DETAILED DESCRIPTION:
Acute lung injury is not uncommon after liver transplantation. A new monitor non-invasive cardiac output monitor (NICOM) is designed to measure thoracic fluid content. The investigators attempt to use the parameter thoracic fluid content to investigate its relationship with acute lung injury in liver transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* end stage liver disease scheduled for liver transplantation in National Taiwna University Hospital.

Exclusion Criteria:

* allergic reaction
* history of aortic regurgitation
* pre-existing pulmonary disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: end stage liver disease patients scheduled for liver transplantation in National Taiwan University Hospital were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2011-01; Primary Completion 2011-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Cardiac index | one day
  Participants will be followed for the duration the operation. Cardiac index was measured by non-invasive cardiac output monitor at different time points as baseline(T1), anhepatic phase(T2), 30 mins after reperfusion(T3) and 2 hrs after reperfusion(T4)

SECONDARY OUTCOMES:
Thoracic fluid content | one day
  Participants will be followed for the duration the operation.Thoracic fluid content was measured in liver transplant recipients at different time points as baseline(T1), anhepatic phase(T2), 30 mins after reperfusion(T3) and 2 hrs after reperfusion(T4).

CONTACTS AND LOCATIONS:
Overall Officials: Kuang Cheng Chan, M.D., Principal Investigator — Department of Anesthesiology, NTUH, Taipei, Taiwan
Locations (1):
- Department of Anesthesiology, NTUH, Taipei, Taiwan

REFERENCES:
- [Background] Hong SK, Hwang S, Lee SG, Lee LS, Ahn CS, Kim KH, Moon DB, Ha TY. Pulmonary complications following adult liver transplantation. Transplant Proc. 2006 Nov;38(9):2979-81. doi: 10.1016/j.transproceed.2006.08.090. PMID 17112879